CLINICAL TRIAL: NCT05208411
Title: The Impact of a Parent-mediated Intervention on Social Behaviour and Social Brain Development in Infants at High Risk for Autism Spectrum Disorder
Brief Title: Prodromal ImPACT Intervention for Children at Elevated Likelihood of ASD
Acronym: SAPIENS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Ghent (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 814302 - ONZ-2022-0587
Record Dates: First submitted 2021-10-20; First posted 2022-01-26 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Autism Spectrum Disorder; Siblings; Preterm; Elevated likelihood of ASD
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Premature Birth

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ImPACT group (Experimental): Group of children at elevated likelihood of ASD who will receive the ImPACT intervention
  Interventions: Behavioral: Project ImPACT: Improving Parents As Communication Teachers
- No intervention group (No Intervention): Group of children at elevated likelihood of ASD who won't receive any intervention

INTERVENTIONS:
Behavioral: Project ImPACT: Improving Parents As Communication Teachers — Project ImPACT ("Improving Parents As Communication Teachers", Ingersoll & Dvortcsak, 2019) is a promising evidence-based parent-mediated intervention that is part of a class of naturalistic, developmental, behavioral interventions (NBDIs). NBDIs involve the use of behavioral principles of learning to teach skills chosen from a developmental sequence in naturalistic play-setting and using natural rewards. Skills selected as relevant for intervention are those that allow the child to participate more fully within reciprocal interactions with the adult. In recent years the program has been adapted for use with infants and toddlers at elevated likelihood of ASD. These adaptations have made this program appropriate for younger children and children who are experiencing social communication delays but do not have an ASD diagnosis.
  Arms: ImPACT group

SUMMARY:
This randomised-controlled trial will assess the effect of an early intervention on the social-communicative abilities and brain activity of infants with elevated likelihood of Autism Spectrum Disorder (ASD). The children´s social-communicative abilities and the related brain activity will be evaluated at three time points: before the start of the intervention (pre-intervention), immediately after its conclusion (post-intervention) and 6 months after its conclusion (follow-up).

DETAILED DESCRIPTION:
Previous research has shown that parent-implemented interventions are effective in improving the social skills of children with autism spectrum disorder (ASD).Considering that several differences in social and non-social skills start to emerge before a diagnosis can be made, this project aims to investigate the effects of an adapted prodromal version of an evidence-based parent-mediated intervention (Project ImPACT) in children with an elevated likelihood to develop ASD (namely siblings and children who were born preterm). The effect of the intervention will be evaluated at both behavioural and neural levels. The intervention is suitable for infants and consists of 12 session with the child and his/her parents, of maximum 2 hours each, one session per week, delivered by therapists of the home guidance and home guidance centers in Flanders. Children between 9 and 18 months old and their parents will participate in the study. They will be randomly assigned to the ImPACT intervention group or a no-intervention group (monitoring only). The families will be invited to come to the Faculty of Psychology and Pedagogical Sciences at three time points: before the start of the intervention, immediately after the end of the intervention (which is expected to last 12 weeks) and 24 weeks after the end of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Elevated likelihood of ASD: the child must be a preterm (less than 30 weeks of gestation) or a sibling/half-sibling of a child with diagnosed ASD.
* Parents are Dutch, English on French speakers.

Exclusion Criteria:

* The child must not have a diagnosis of other neurological or developmental disorders.

Ages: 9 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 80 (Estimated)
Dates: Start 2022-03-28 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Bigger change from baseline in the parent-child interaction in the intervention group compared to the no-intervention group. | Outcome at 3 months after entry(post-test)
  Change in quality and frequency of behaviours (with the same unit of measure) within the Parent-Child Interaction coded through the Parent-Infant/Toddler Coding of Interaction (PInTCI). An increase is considered as a positive outcome.
Bigger change from post-test in the intervention group in the parent-child interaction compared to the no-intervention group. | Follow-up at 6 months after post-test
  Change in quality and frequency of behaviours (with the same unit of measure) within the Parent-Child Interaction coded through the Parent-Infant/Toddler Coding of Interaction (PInTCI). An increase is considered as a positive outcome.

SECONDARY OUTCOMES:
Bigger change from baseline in Social Engagement in the intervention group compared to the no-intervention group. | outcome at 3 months after entry (post-test)
  Duration of the engagement in interactive play with the adult. Consider whether the child 1) engages in interactive play, 2) follows the adult's lead in play activities; 3) sustains interactive play (e.g. by requesting for the activity to continue) and 4) initiates the adults engagement in interactive play. The total Social Engagement score will consist of a composite score of the abovementioned aspects coded during the administration of both the Communication and Symbolic Behavior Scale (CSBS) and the Early Social Communication Scales (ESCS).
  Higher frequency and longer social engagement time is considered positive outcome.
Bigger change from baseline in the score of imitation in the intervention group compared to the no-intervention group. | outcome at 3 months after entry (post-test)
  Semi-structured social imitation task developed by B. Ingersoll, author of the ImPACT intervention programme. Semi-structured observation of interaction with experimenter. Only the object scale is used. The score ranges from 0 to 20, with higher scores corresponding to higher social imitation rates.
  Score increase is a positive outcome.
Bigger change from baseline in the score of intentional communication in the intervention group compared to the no-intervention group | outcome at 3 months after entry (post-test)
  Composite weighted frequency of unprompted intentional triadic communication (initiations), obtained by multiplying each unprompted triadic communication act by the weight assigned to the behaviour used to communicate. The total Intentional Communication score will consist of a composite score of the abovementioned aspects coded during the administration of both the Communication and Symbolic Behavior Scale (CSBS) and the Early Social Communication Scales (ESCS).
  Score increase is a positive outcome.
Bigger change from baseline in attention disengagement in the intervention group compared to the no-intervention group | outcome at 3 months after entry (post-test)
  Attention disengagement is defined as the time needed to shift the gaze to a peripheral target. It's measured with an Eye-tracker while presenting a well-known paradigm called Gap-Overlap task.
  Decrease in Attention disengagement time is considered as a positive outcome.
Bigger change from baseline in the intervention group compared to the no-intervention group in electrophysiological spectral power and connectivity (theta and alpha band) in response to social versus non-social videos, measured with EEG. | outcome at 3 months after entry (post-test)
  EEG activity recorded while children watch videos of abstract figures moving (resting-state), social scenes (nursery rhymes) and non-social scenes (toys moving).
Bigger change from post-test in the intervention group in the score of Social Engagement compared to the no-intervention group. | follow-up at 6 months after post-test
  Duration of the engagement in interactive play with the adult. Consider whether the child 1) engages in interactive play, 2) follows the adult's lead in play activities; 3) sustains interactive play (e.g. by requesting for the activity to continue) and 4) initiates the adults engagement in interactive play. The total Social Engagement score will consist of a composite score of the abovementioned aspects coded during the administration of both the Communication and Symbolic Behavior Scale (CSBS) and the Early Social Communication Scales (ESCS). Score stability (after increase at outcome) or increase is a positive outcome.
Bigger change from post-test in the score of a semi-structured social imitation task compared to the no-intervention group. | follow-up at 6 months after post-test
  Semi-structured social imitation task developed by B. Ingersoll, author of the ImPACT intervention programme. Semi-structured observation of interaction with experimenter. Only the object scale is used. The score ranges from 0 to 20, with higher scores corresponding to higher social imitation rates.
  Score stability (after increase at outcome) or increase is a positive outcome.
Bigger change from post-test in the score of intentional communication in the intervention group compared to the no-intervention group | follow-up at 6 months after post-test
  Composite weighted frequency of unprompted intentional triadic communication (initiations), obtained by multiplying each unprompted triadic communication act by the weight assigned to the behaviour used to communicate. The total Intentional Communication score will consist of a composite score of the abovementioned aspects coded during the administration of both the Communication and Symbolic Behavior Scale (CSBS) and the Early Social Communication Scales (ESCS). Score stability (after increase at outcome) or increase is a positive outcome.
Bigger change from post-test in the intervention group in electrophysiological spectral power and connectivity (theta and alpha band) in response to social versus non-social videos, measured with EEG. | follow-up at 6 months after post-test
  EEG activity recorded while children watch videos of abstract figures moving (resting-state), social scenes (nursery rhymes) and non-social scenes (toys moving).
Bigger change from post-test in attention disengagement in the intervention group compared to the no-intervention group, measured with Eye-tracking | follow-up at 6 months after post-test
  Attention disengagement is the time needed to shift the gaze to a peripheral target. It's measured with an Eye-tracker while presenting a well-known paradigm called Gap-Overlap task.
  Attention disengagement time stability (after decrease at outcome) or decrease is a positive outcome.
Difference between intervention and no-intervention group in the severity score of the Autism Diagnostic Observational Scale - 2 (ADOS-2). | outcome at 9 months after entry
  A standard measure internationally used to identify symptoms of autism. The total score ranges from 0 to 30, with a higher score corresponding to higher symptom severity. The total score results from the sum of two subscales: the Social Affect subscale (SA), with scores ranging from 0 to 22, and the Restricted and Repetitive Behavior one (RRB), with scores ranging from 0 to 8. The ADOS-2 total score is converted through an age-dependent algorithm to a diagnostic ordinal scale ranging from 0 to 10 (with higher scores indicating higher symptom severity), based on which a diagnostic classification can be formulated (no ASD, ASD, autism).
  A lower total score in the intervention group, as well as in a subscale score, compared to the no-intervention group is considered a positive outcome.
Bigger change from baseline in the in the intervention group in the score of the Bayley Scales of Infant and Toddler Development - Third Edition - NL compared to the no-intervention group. | outcome at 9 months after entry
  An age-appropriate measure of cognitive, language, motor and social-emotional development for children from 0 to 42 months. A high growth rate (= the change in months is higher than the number of months actually passed between baseline and follow-up) in a domain where a child initially showed a delay is considered a positive outcome.
Bigger change from baseline in the intervention group score of the Nijmeegse Ouderlijke Stress Index compared to the no-intervention group. | outcome at 9 months after entry
  Questionnaire over Parenting stress index developed in Nijmegen. Scores range from 0 to 738, distributed over two main subscales: parent-related stress and child-related stress. Each subscale is composed of subdomains. The parent-related stress is described by competence, role restriction, attachment, depression, health, social isolation, marital relationship. The child-related stress is described by adaptation, temperament, distractibility, demandingness, positive reinforcement, acceptance. An algorithm converts the subscores and the total score to a descriptive classification of parental stress level. Special norms hold for clinical samples.
  Higher values correspond to higher parental stress. A score reduction is a positive outcome, in particular if lower than the no-intervention group.
Bigger change from baseline in the intervention group score of the Vineland screener questionnaire (0-6 years) compared to the no-intervention group. | outcome at 9 months after entry
  Questionnaire to assess adaptive skills. The composite score is computed as the sum of subscale scores: communicative skills (0-38), social skills (0-38), everyday skills (0-16), motor skills (0-36). Raw scores can be converted to adaptive age.
  Score stability (after increase) or increase is a positive outcome, in particular if higher than the no-intervention group.
Difference between intervention and no-intervention group in language. | outcome at 9 months after entry
  Language will be investigated with the Dutch adaptation of the MacArthur Communicative Development Inventories (CDI), Words and Gestures (8-18 months) and Words and Sentences (16-30 months), which consists of a parent report of language development (both comprehension and production).
  Higher score in the intervention group is considered a positive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. Herbert Roeyers, PhD, Study Chair — University Ghent
Locations (1):
- Ghent University, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No